CLINICAL TRIAL: NCT03178188
Title: Efficacy of 595 nm Pulsed-dye Laser as an Adjunctive Treatment of Discoid Lupus Erythematosus, A Randomized, Patient/Assessor Blinded Placebo Control Trial
Brief Title: Efficacy of 595 nm Pulsed-dye Laser in Treatment of Discoid Lupus Erythematosus
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Pawinee Rerknimitr, Assistant Professor, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1/59
Record Dates: First submitted 2017-06-02; First posted 2017-06-06 (Actual); Last update posted 2017-06-06 (Actual); Status verified 2017-06

CONDITIONS: Lupus Erythematosus, Discoid
Keywords: lupus erythematosus, Discoid; Pulsed-dye Laser
MeSH Terms: conditions — Lupus Erythematosus, Discoid | interventions — Lasers, Dye

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- laser treated DLE lesions (Experimental): DLE which received the pulsed-dye laser
  Interventions: Device: Pulsed-dye Laser
- sham treated DLE lesions (Sham Comparator): DLE which received the sham
  Interventions: Device: Sham

INTERVENTIONS:
Device: Pulsed-dye Laser — 595 nm Pulsed-dye Laser; 7mm spot sizes, 6msec pulse durations, 8j/cm2 fluences, dynamic cooling device 30/20, 4 sessions with 4 weeks interval
  Arms: laser treated DLE lesions
Device: Sham — Cryogen spray with the setting of dynamic cooling device 30/20
  Arms: sham treated DLE lesions

SUMMARY:
forty DLE lesions from patients will be recruited in the study. The lesions on one side of the body were block-randomized into the treatment group and the other side served as a control. The patients can continue their systemic treatments and the PDL is designed to be used as an adjunctive treatment. Treatments with the PDL will be delivered in the treatment group every 4 weeks for 4 consecutive months while the lesions in the control group received a sham. The patients will be evaluated at baseline (week 0), week 4, 8, 12, and at follow-up period of 4, 12 weeks after the final treatment (week 16, 24). Erythema index (EI), Texture index (TI) will be obtained and digital photographs will be taken and modified Cutaneous Lupus Erythematosus Disease Area and Severity Index (mCLASI) will be assessed in every visit. The digital photographs will later be evaluated by 3-blinded dermatologists. Moreover, side effects and patients' satisfaction score will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Has at least two DLE lesions, located in the same anatomical location of the body, which the different of mCLASI are not more than 1 point
* Dose not undergo any procedure or laser treatment within 4 weeks before entered the study
* Dose not received any localised therapy of DLE eg. topical corticosteriod/immunomodulator within 4 weeks before entered the study
* Dose not receive the topical chemical peeling within 4 weeks before entered the study
* Has already received at least 1 systemic standard treatment for DLE and continue until the rest of the study
* Can follow the study's protocol

Exclusion Criteria:

* Pregnancy or lactation
* History of skin cancer
* History of photo allergy
* History of bleeding tendency
* History of abnormal wound healing

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2016-12-15 (Actual); Primary Completion 2017-12-14 (Estimated); Study Completion 2017-12-14 (Estimated)

PRIMARY OUTCOMES:
erythema index (EI) | week 0(baseline), 4, 8, 12, 16, 24
  Comparing changes of EI from baseline between treated group and controlled group, measured by Antera 3D camera

SECONDARY OUTCOMES:
modified Cutaneous Lupus Erythematosus Disease Area and Severity Index(mCLASI) | week 0, 4, 8, 12, 16, 24
  Comparing changes of mCLASI from baseline between treated group and controlled group, measured by 1-blinded dermatologist
Physician Global Assessment (PGA) scores | week 0, 4, 8, 12, 16, 24
  Comparing overall improvement changes from baseline (PGA scores) measured by 3-blinded dermatologist
texture index (TI) | week 0, 4, 8, 12, 16, 24
  Comparing changes of TI from baseline between treated group and controlled group, measured by Antera 3D camera

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Dermatology, Faculty of Medicine, Chulalongkorn University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No